CLINICAL TRIAL: NCT06547801
Title: Effects of Human Milk Oligosaccharide Ingestion on Weight Loss and Markers of Health
Acronym: HMO-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Protein Technologies Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB2022-1559F; APT00001 (Other Grant/Funding Number: Advanced Protein Technologies Corp.)
Record Dates: First submitted 2024-06-11; First posted 2024-08-09 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Weight Loss
Keywords: 2'-Fucosyllactose; Inflammation; Functional capacity
MeSH Terms: conditions — Weight Loss; Inflammation | interventions — 2'-fucosyllactose; maltodextrin

STUDY DESIGN:
Intervention Model Description: This study was conducted as a randomized, double-blind, placebo-controlled, parallel arm study. The Human Protection Institutional Review Board (IRB2022-1559F) approved the study following ethical standards for the conduct of human participant research as described in the Declaration of Helsinki.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2'-fucosyllactose (Experimental): 3 g/day of 2'-FL powder orally once daily for 12 weeks
  Interventions: Dietary Supplement: 2'-Fucosyllactose
- Maltodextrin (Placebo Comparator): 3 g/day of banana-flavored maltodextrin powder orally once daily for 12 weeks
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: 2'-Fucosyllactose — 3 g/day of powder orally once daily
  Arms: 2'-fucosyllactose
Dietary Supplement: Maltodextrin — 3 g/day of powder orally once daily
  Arms: Maltodextrin

SUMMARY:
A randomized, double-blind, placebo-controlled, parallel arm study of 2'-fucosyllactose (2'-FL) was conducted in healthy males and females between the ages of 18 and 65 at the time of consent. 2'-FL is one of the most prominent HMOs in human milk. Preclinical studies indicate that 2'-FL feeding is prebiotic, anti-inflammatory, anti-thrombotic, and may reduce skeletal muscle atrophy during energy restriction. The investigators hypothesize that supplementation of 2'-FL affects the preservation of muscle mass, strength, and markers of health during exercise and a hypo-energetic weight loss program. To test this hypothesis, the investigators will compare 3 g/day of 2'-FL with 3 g/day of maltodextrin placebo as a daily supplement.

DETAILED DESCRIPTION:
Objective: To investigate the effects of daily supplementation with 3 g/day of 2'-fucosyllactose (2'-FL) compared to 3 g/day of maltodextrin placebo on muscle mass preservation, strength, and health markers during exercise and a hypo-energetic weight loss program in healthy adults.

Study Design: This study will be a randomized, double-blind, placebo-controlled, parallel arm trial.

Participants: Participants will include healthy males and females aged 18 to 65 years at the time of consent, with a BMI between 25 to 40 kg/m² and/or body fat greater than 30%. Preference will be given to individuals with a BMI between 25 to 32 kg/m² who express a desire to lose weight and participate in a fitness exercise program.

Intervention: Participants will be randomly assigned to receive either 3 g/day of 2'-FL or 3 g/day of maltodextrin placebo, administered daily for the duration of the study.

Ethical Considerations: This study will adhere to ethical guidelines for human research, ensuring participant confidentiality, informed consent, and data protection.

Timeline: The study will commence upon institutional approval and is expected to be completed within 12 weeks.

This study aims to provide insights into the potential benefits of 2'-FL supplementation on muscle preservation, strength, and overall health during exercise and weight loss efforts, contributing to the understanding of its role as a dietary supplement.

ELIGIBILITY:
Inclusion Criteria:

* Men and women the ages of 18 to 65 at the time of consent
* Ability to comply with study procedures
* Availability to complete the study based on duration of individual visits and scheduling requirements
* Body mass index (BMI) between 25 and 40 kg/m2 and/or body fat less than 30%, with a preference between a BMI of 25 - 32 kg/m2, and a desire to lose weight and participate in a fitness exercise program

Exclusion Criteria:

* Pregnant, breastfeeding, or wish to become pregnant during the study
* Planning major changes in lifestyle (i.e., diet, dieting, exercise level, travel) during the study
* Recent history (< 3 months) of exercise training or weight loss (> 5%)
* Orthopedic limitation preventing participation in a general fitness program
* Uncontrolled heart disease, hypertension, diabetes, thyroid disease, cancer, neurological disease, or untreated psychotic or major depressive disorder in which participation in a general fitness program is contraindicated
* Taking weight loss dietary supplements or medications during the last 4 weeks
* History within the previous 12 months of alcohol or substance abuse
* Heavy smoking (> 1 pack/day within the past 3 months)
* Known allergy to milk, lactose, or any other milk product

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Change in Body Weight | baseline (0 weeks), midpoint (6 weeks), and endpoint (12 weeks)
  Change in body weight (kilograms) using a calibrated digital scale
Change in Body Height | baseline (0 weeks), midpoint (6 weeks), and endpoint (12 weeks)
  Change in height (meters) using a calibrated digital scale
Change in Body Mass Index (BMI) | baseline (0 weeks), midpoint (6 weeks), and endpoint (12 weeks)
  Body Mass Index (BMI) calculated using weight and height, expressed in kg/m².
Change in Fat Mass | baseline (0 weeks), midpoint (6 weeks), and endpoint (12 weeks)
  Change in fat mass (kilograms) measured using a calibrated Hologic Discovery W (Hologic Inc., Waltham, MA, USA) with APEX Software (APEX Corporation, Pittsburgh, PA, USA).
Change in Lean Body Mass | baseline (0 weeks), midpoint (6 weeks), and endpoint (12 weeks)
  Lean body mass (kilograms) calculated using Hologic Discovery W (Hologic Inc., Waltham, MA, USA) with APEX Software (APEX Corporation, Pittsburgh, PA, USA).
Change in Body Fat | baseline (0 weeks), midpoint (6 weeks), and endpoint (12 weeks)
  Body fat percentage calculated using Hologic Discovery W (Hologic Inc., Waltham, MA, USA) with APEX Software (APEX Corporation, Pittsburgh, PA, USA).
Change in Bone Mineral Content | baseline (0 weeks), midpoint (6 weeks), and endpoint (12 weeks)
  Bone mineral content (grams) measured using Hologic Discovery W (Hologic Inc., Waltham, MA, USA) with APEX Software (APEX Corporation, Pittsburgh, PA, USA).
Change in Waist Circumference | baseline (0 weeks), midpoint (6 weeks), and endpoint (12 weeks)
  Waist circumference (centimeters) measured with a soft tape.
Change in Hip Circumference | baseline (0 weeks), midpoint (6 weeks), and endpoint (12 weeks)
  Hip circumference (centimeters) measured with a soft tape.

SECONDARY OUTCOMES:
Change in Aerobic Capacity | baseline (0 weeks), midpoint (6 weeks), and endpoint (12 weeks)
  Change in peak oxygen uptake (L/min) from baseline.
Change in White Blood cell | baseline (0 weeks), midpoint (6 weeks), and endpoint (12 weeks)
  White Blood cells (K/uL) were analyzed from collected fasting whole blood samples.
Change in Red Blood cell | baseline (0 weeks), midpoint (6 weeks), and endpoint (12 weeks)
  Red Blood cells (M/uL) were analyzed from collected fasting whole blood samples.
Change in Hemoglobin | baseline (0 weeks), midpoint (6 weeks), and endpoint (12 weeks)
  Hemoglobins (g/dL) were analyzed from collected fasting whole blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Kreider, Professor, Study Director — rbkreider@tamu.edu
Locations (1):
- Exercise & Sport Nutrition Lab, Department of Kinesiology and Sport Management, Texas A&M University, College Station, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pak ME, Kim YJ, Kim H, Shin CS, Yoon JW, Jeon SM, Song YH, Kim K. Anti-Neuroinflammatory Effects of the Human Milk Oligosaccharide, 2'-Fucosyllactose, Exerted via Modulation of M2 Microglial Activation in a Mouse Model of Ischemia-Reperfusion Injury. Antioxidants (Basel). 2023 Jun 15;12(6):1281. doi: 10.3390/antiox12061281. PMID 37372011
- [Background] Le Huerou-Luron I, Blat S, Boudry G. Breast- v. formula-feeding: impacts on the digestive tract and immediate and long-term health effects. Nutr Res Rev. 2010 Jun;23(1):23-36. doi: 10.1017/S0954422410000065. Epub 2010 May 10. PMID 20450531
- [Background] Ikeda N, Shoji H, Murano Y, Mori M, Matsunaga N, Suganuma H, Ikeno M, Hisata K, Hirayama S, Ueno T, Miida T, Shimizu T. Effects of breastfeeding on the risk factors for metabolic syndrome in preterm infants. J Dev Orig Health Dis. 2014 Dec;5(6):459-64. doi: 10.1017/S2040174414000397. Epub 2014 Aug 28. PMID 25167084
- [Background] Saarinen UM, Kajosaari M. Breastfeeding as prophylaxis against atopic disease: prospective follow-up study until 17 years old. Lancet. 1995 Oct 21;346(8982):1065-9. doi: 10.1016/s0140-6736(95)91742-x. PMID 7564787
- [Result] Elison E, Vigsnaes LK, Rindom Krogsgaard L, Rasmussen J, Sorensen N, McConnell B, Hennet T, Sommer MO, Bytzer P. Oral supplementation of healthy adults with 2'-O-fucosyllactose and lacto-N-neotetraose is well tolerated and shifts the intestinal microbiota. Br J Nutr. 2016 Oct;116(8):1356-1368. doi: 10.1017/S0007114516003354. Epub 2016 Oct 10. PMID 27719686
- [Result] Vazquez E, Barranco A, Ramirez M, Gruart A, Delgado-Garcia JM, Jimenez ML, Buck R, Rueda R. Dietary 2'-Fucosyllactose Enhances Operant Conditioning and Long-Term Potentiation via Gut-Brain Communication through the Vagus Nerve in Rodents. PLoS One. 2016 Nov 16;11(11):e0166070. doi: 10.1371/journal.pone.0166070. eCollection 2016. PMID 27851789
- [Result] Teixeira V, Voci SM, Mendes-Netto RS, da Silva DG. The relative validity of a food record using the smartphone application MyFitnessPal. Nutr Diet. 2018 Apr;75(2):219-225. doi: 10.1111/1747-0080.12401. Epub 2017 Dec 27. PMID 29280547
- [Result] Thompson PD, Arena R, Riebe D, Pescatello LS; American College of Sports Medicine. ACSM's new preparticipation health screening recommendations from ACSM's guidelines for exercise testing and prescription, ninth edition. Curr Sports Med Rep. 2013 Jul-Aug;12(4):215-7. doi: 10.1249/JSR.0b013e31829a68cf. No abstract available. PMID 23851406
- [Result] Nishida C, Ko GT, Kumanyika S. Body fat distribution and noncommunicable diseases in populations: overview of the 2008 WHO Expert Consultation on Waist Circumference and Waist-Hip Ratio. Eur J Clin Nutr. 2010 Jan;64(1):2-5. doi: 10.1038/ejcn.2009.139. Epub 2009 Nov 25. PMID 19935820
- [Result] Lohman TG, Harris M, Teixeira PJ, Weiss L. Assessing body composition and changes in body composition. Another look at dual-energy X-ray absorptiometry. Ann N Y Acad Sci. 2000 May;904:45-54. doi: 10.1111/j.1749-6632.2000.tb06420.x. PMID 10865709
- [Result] Klesges RC, Ward KD, Shelton ML, Applegate WB, Cantler ED, Palmieri GM, Harmon K, Davis J. Changes in bone mineral content in male athletes. Mechanisms of action and intervention effects. JAMA. 1996 Jul 17;276(3):226-30. PMID 8667568
- [Result] Peronnet F, Massicotte D. Table of nonprotein respiratory quotient: an update. Can J Sport Sci. 1991 Mar;16(1):23-9. PMID 1645211
- [Result] Gupta RD, Ramachandran R, Venkatesan P, Anoop S, Joseph M, Thomas N. Indirect Calorimetry: From Bench to Bedside. Indian J Endocrinol Metab. 2017 Jul-Aug;21(4):594-599. doi: 10.4103/ijem.IJEM_484_16. PMID 28670546
- [Result] Page P. Beyond statistical significance: clinical interpretation of rehabilitation research literature. Int J Sports Phys Ther. 2014 Oct;9(5):726-36. PMID 25328834
- [Derived] Ko J, Yoo C, Xing D, Chun J, Gonzalez DE, Dickerson BL, Leonard M, Jenkins V, van der Merwe M, Slupsky CM, Sowinski R, Rasmussen CJ, Kreider RB. Effects of Human Milk Oligosaccharide 2'-Fucosyllactose Ingestion on Weight Loss and Markers of Health. Nutrients. 2024 Oct 5;16(19):3387. doi: 10.3390/nu16193387. PMID 39408354